CLINICAL TRIAL: NCT00757913
Title: The Effect of n-3 Enriched Nutrition Therapy on Postoperative Cognitive Dysfunction and Delirium After Elective Cardiac Surgery
Brief Title: n-3 Enriched Nutrition Therapy and Postoperative Cognitive Dysfunction After Cardiac Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment rate
Sponsor: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EK 92/08
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Delirium, Dementia, Amnestic, Cognitive Disorders; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Neurocognitive Disorders; Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): n-3 enriched nutrition
  Interventions: Dietary Supplement: n-3 enriched nutrition
- 2 (Placebo Comparator): isocaloric nutrition without n-3 supplement
  Interventions: Dietary Supplement: n-3 enriched nutrition

INTERVENTIONS:
Dietary Supplement: n-3 enriched nutrition

SUMMARY:
Background: Delirium and long-term cognitive dysfunction (CD) are important complications of major surgery and intensive care treatment. Delirium is associated with increased mortality and CD has an important impact on mortality, independency, social interactions, and quality of life. Delirium is an important risk factor for the development of long-term CD. Particularly, patients aged 65 or older undergoing cardiac surgery are at a high risk of developing these problems. There are data suggesting that inflammation plays a key role in the development of delirium and possibly CD. It has been shown that n-3 fatty acids modulate the immune response of patients and have beneficial effects in abdominal surgery.

Working hypothesis: 1. Administration of n-3 enriched nutrition therapy including will modulate the inflammatory response and improve cognitive function after cardiac surgery.

Specific Aims: This project will test the impact of perioperative enteral n-3 fatty acids ProSure, Abbott Nutrition) in elderly patients undergoing elective cardiac surgery. Primary endpoint is CD one week postoperatively.

Methods: The investigators will investigate 400 patients aged 65 or older undergoing elective cardiac surgery. Half of these patients will receive supplementary of n-3 fatty acids to modulate the inflammatory response; the other half will receive an isocaloric nutritional supplement without n-3 fatty acids (Ensure Plus, Abbott Nutrition). Otherwise the treatment of the patients will not be influenced by this study. Cognitive function will be assessed preoperatively, 7 days and three months postoperatively. C-reactive protein, IL-6, IL-8, IL-10, S-100B, and neuron specific enolase will be monitored as markers of systemic inflammation and delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patient's undergoing elective cardiac procedure with extracorporeal circulation
* Age 65 or older

Exclusion Criteria:

* No informed written consent
* "Redo" operation
* Deep hypothermic cardiac arrest
* Operation including carotid endarterectomy
* Known allergy to n-3 fatty acids
* History of cerebrovascular disease
* Preoperative Mini mental score < 23
* Long term neuroleptic medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative cognitive dysfunction 7 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Luzius A Steiner, MD, PhD, Principal Investigator — Department of Anaesthesia, University Hospital Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland